CLINICAL TRIAL: NCT00098293
Title: A Multicenter, Randomized, Double-Blind, Comparative Trial Of A Novel CCR5 Antagonist, UK-427,857, In Combination With Zidovudine/Lamivudine Versus Efavirenz In Combination With Zidovudine/Lamivudine For The Treatment Of Antiretroviral-Naive HIV-1 Infected Subjects
Brief Title: Trial of Maraviroc (UK-427,857) in Combination With Zidovudine/Lamivudine Versus Efavirenz in Combination With Zidovudine/Lamivudine
Acronym: MERIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4001026
Record Dates: First submitted 2004-12-06; First posted 2004-12-07 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-08

CONDITIONS: HIV-1
Keywords: Aids; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Zidovudine; Lamivudine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Maraviroc + Zidovudine/Lamivudine
- 3 (Active Comparator)
  Interventions: Drug: Efavirenz + Zidovudine/Lamivudine
- 2 (Experimental): Following a review of the interim analysis data, the DSMB recommended to terminate the UK-427,857 300 mg QD arm based on pre-specified protocol non-inferiority criteria not being met for the QD arm versus efavirenz
  Interventions: Drug: Maraviroc (UK-427,857) + Zidovudine/Lamivudine

INTERVENTIONS:
Drug: Maraviroc + Zidovudine/Lamivudine — maraviroc (UK-427,857) 300 mg once daily added to zidovudine/lamivudine (300 mg/150 mg twice daily)
  Arms: 1
Drug: Efavirenz + Zidovudine/Lamivudine — efavirenz (600 mg once daily) added to zidovudine/lamivudine (300 mg/150 mg twice daily)
  Arms: 3
Drug: Maraviroc (UK-427,857) + Zidovudine/Lamivudine — maraviroc (UK-427,857) 300 mg twice daily added to zidovudine/lamivudine (300 mg/150 mg twice daily)
  Arms: 2

SUMMARY:
Maraviroc (UK-427,857), a selective and reversible CCR5 coreceptor antagonist, has been shown to be active in vitro against a wide range of clinical isolates (including those resistant to existing classes). In HIV-1 infected patients, maraviroc (UK-427,857) given as monotherapy for 10 days reduced HIV-1 viral load by up to 1.6 log, consistent with currently available agents. Safety and toleration have been studied in over 400 subjects for up to 28 days at 300 mg twice daily. No significant effects were seen on the QTc interval. The goal of this study is to compare the safety and efficacy of maraviroc (UK-427,857) versus efavirenz, when each are combined with two other antiretroviral agents, in patients who are previously naive to antiretroviral therapy. This study will involve approximately 200 centers from around the world to achieve a total randomized subject population of 1071 subjects. Patients will be randomly assigned to one of three groups: maraviroc (UK-427,857) 300 mg once daily added to zidovudine/lamivudine (300 mg/150 mg twice daily), Maraviroc (UK-427,857) 300 mg twice daily added to zidovudine/lamivudine (300 mg/150 mg twice daily) or efavirenz (600 mg once daily) added to zidovudine/lamivudine (300 mg/150 mg twice daily). The study will enroll over approximately an 18 month period (5 months Phase 2b run-in, 13 months Phase 3) with 96 weeks of treatment. This may be extended for an additional 3 years depending on the results at 96 weeks. Physical examinations will be performed at study entry, weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96. Blood samples will also be taken at study entry, weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, 60, 72, 84 and 96. Additionally, blood samples will be drawn twice, at least 30 minutes apart, at weeks 2 and 48 for maraviroc (UK-427,857) pharmacokinetic analysis. As part of this clinical study a blood sample will be taken for non-anonymized pharmacogenetic analysis. Patients will undergo a 12-lead electrocardiogram at study entry, weeks 24, 48 and 96. A computerized tomography (CT) scan will also be performed, at selected centers, at study entry and week 96. Patients will be asked to complete a symptom distress questionnaire at study entry, weeks 12, 24, 48 and 96.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 16 years of age (or minimum age as determined by local regulatory authorities)
* HIV-1 RNA viral load of greater than or equal to 2, 000 copies/mL
* A negative urine pregnancy test at the baseline visit for Women of Child Bearing Potential (WOCBP)
* Effective barrier contraception for WOCBP and males

Exclusion Criteria:

* Suspected or documented active, untreated HIV-1 related opportunistic infection (OI) or other condition requiring acute therapy
* Treatment for an active opportunistic infection, or unexplained temperature >38.5 degrees Celsius for 7 consecutive days
* Prior treatment with efavirenz, zidovudine or lamivudine or with any other antiretroviral therapy for more than 14 days at any time
* Active alcohol or substance abuse sufficient, in the Investigator's judgment, to prevent adherence to study medication and/or follow up
* Lactating women, or planned pregnancy during the trial period
* Suspected primary (acute) HIV-1 infection
* Previous therapy with a potentially myelosuppressive, neurotoxic, hepatotoxic and/or cytotoxic agent within 30 days prior to randomization or the expected need for such therapy during the study period
* Documented or suspected acute hepatitis or pancreatitis within 30 days prior to randomization
* Significantly elevated liver enzymes or cirrhosis
* Significant neutropenia, anemia or thrombocytopenia
* Malabsorption or an inability to tolerate oral medications
* Symptomatic postural hypotension or severe cardiovascular or cerebrovascular disease
* Certain medications
* Genotypic or phenotypic resistance to efavirenz, zidovudine or lamivudine
* X4- or dual/mixed-tropic virus or repeated assay failure
* Any other clinical condition that, in the Investigator's judgement, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 916 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (111):
- United States (36):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Flushing, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Argentina (7):
  - Pfizer Investigational Site, El Palomar, Buenos Aires
  - Pfizer Investigational Site, Neuquén, Neuquén Province
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Ciudad de Buenos Aires
  - Pfizer Investigational Site, Ciudad de Buenos
  - Pfizer Investigational Site, Provincia de Buenos Aires
  - Pfizer Investigational Site, Provincia de Santa Fe
- Australia (9):
  - Pfizer Investigational Site, Burwood, New South Wales
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Surrey Hills, New South Wales
  - Pfizer Investigational Site, Wentworthville, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Miami, Queensland
  - Pfizer Investigational Site, Fitzroy North, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, South Yarra, Victoria
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (10):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
- Italy (6):
  - Pfizer Investigational Site, Antella (FI)
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Modena
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Torino
- Mexico (3):
  - Pfizer Investigational Site, Del. Tlalpan C.P., Mexico City
  - Pfizer Investigational Site, Del. Tlalpan, C.P., Mexico City
  - Pfizer Investigational Site, Delegacion Tlalpan C. P, Mexico City
- Netherlands (3):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Utrecht
- Poland (7):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Chorzów
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Puerto Rico (3):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, Rio Piedras
  - Pfizer Investigational Site, San Juan
- South Africa (11):
  - Pfizer Investigational Site, Port Elizabeth, Eastern Cape
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Dundee, KwaZulu-Natal
  - Pfizer Investigational Site, Bloomfontein
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Pretoria North
  - Pfizer Investigational Site, Soweto, Johannesburg
- Switzerland (6):
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
  - Pfizer Investigational Site, Lugano
  - Pfizer Investigational Site, Sankt Gallen
  - Pfizer Investigational Site, Zurich
- United Kingdom (6):
  - Pfizer Investigational Site, Edinburgh, Loth
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Brighton
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Vourvahis M, McFadyen L, Nepal S, Valluri SR, Fang A, Fate GD, Wood LS, Marshall JC, Chan PLS, Nedderman A, Haynes J, Savage ME, Clark A, Smith KY, Heera J. No Clinical Impact of CYP3A5 Gene Polymorphisms on the Pharmacokinetics and/or Efficacy of Maraviroc in Healthy Volunteers and HIV-1-Infected Subjects. J Clin Pharmacol. 2019 Jan;59(1):139-152. doi: 10.1002/jcph.1306. Epub 2018 Sep 7. PMID 30192390
- [Derived] MacInnes A, Lazzarin A, Di Perri G, Sierra-Madero JG, Aberg J, Heera J, Rajicic N, Goodrich J, Mayer H, Valdez H. Maraviroc can improve lipid profiles in dyslipidemic patients with HIV: results from the MERIT trial. HIV Clin Trials. 2011 Jan-Feb;12(1):24-36. doi: 10.1310/hct1201-24. PMID 21388938
- [Derived] Funderburg N, Kalinowska M, Eason J, Goodrich J, Heera J, Mayer H, Rajicic N, Valdez H, Lederman MM. Effects of maraviroc and efavirenz on markers of immune activation and inflammation and associations with CD4+ cell rises in HIV-infected patients. PLoS One. 2010 Oct 6;5(10):e13188. doi: 10.1371/journal.pone.0013188. PMID 20949133
- [Derived] Cooper DA, Heera J, Goodrich J, Tawadrous M, Saag M, Dejesus E, Clumeck N, Walmsley S, Ting N, Coakley E, Reeves JD, Reyes-Teran G, Westby M, Van Der Ryst E, Ive P, Mohapi L, Mingrone H, Horban A, Hackman F, Sullivan J, Mayer H. Maraviroc versus efavirenz, both in combination with zidovudine-lamivudine, for the treatment of antiretroviral-naive subjects with CCR5-tropic HIV-1 infection. J Infect Dis. 2010 Mar 15;201(6):803-13. doi: 10.1086/650697. PMID 20151839
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001026&StudyName=Trial%20of%20Maraviroc%20%28UK-427%2C857%29%20in%20Combination%20with%20Zidovudine/Lamivudine%20versus%20Efavirenz%20in%20Combination%20with%20Zidovudine/Lamivudine

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data Safety Monitoring Board (DSMB) recommended termination of maraviroc once daily treatment after interim analysis at nominal week 16, 130 participants of 177 randomized were switched to open-label (OL) maraviroc twice daily.
Groups:
- Maraviroc Once Daily + CBV (DB): Maraviroc 300 milligram (mg) tablet orally once daily in the evening along with placebo matched to maraviroc 300 mg tablet orally once daily in the morning and placebo matched to efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the double-blind (DB) phase prior to the termination of the treatment arm based on the recommendation of the DSMB following a planned interim analysis. DB phase nominally ended at last participant's Week 96 visit.
- Maraviroc Twice Daily + CBV (DB and OL): Maraviroc 300 mg tablet orally twice daily and placebo matched to efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the DB phase. DB phase nominally ended at last participant's Week 96 visit. Maraviroc 300 mg tablet orally twice daily co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the open-label (OL) phase. OL phase continued for at least 3 years after DB phase.
- Efavirenz Once Daily + CBV (DB and OL): Placebo matched to maraviroc 300 mg tablet orally twice daily and efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the DB phase. DB phase nominally ended at last participant's Week 96 visit. Efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the OL phase. OL phase continued for at least 3 years after DB phase.
- Maraviroc Twice Daily + CBV (OL): Participants who received maraviroc 300 mg tablet orally once daily treatment during the DB phase and who were eligible based on safety criteria and virologic response, switched to OL maraviroc 300 mg tablet orally twice daily co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, following the DSMB recommendation to terminate the maraviroc once daily treatment arm after planned interim analysis. OL phase continued for at least 3 years after DB phase.
- Maraviroc Twice Daily + CBV (SP): Participants who remained on mararviroc until their open-label phase End-of-Study visit and for whom maraviroc was commercially or otherwise unavailable entered an additional supplemental phase (SP) (initially planned for 6 months and subsequently extended for another 6 months) which consisted of study visits at 3-month intervals and received maraviroc 300 mg tablet orally twice daily co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily until maraviroc was commercially or otherwise available.
Period: Double-blind (DB) Phase
Arm/Group | Maraviroc Once Daily + CBV (DB) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Maraviroc Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (SP)
Started | 177 | 368 | 372 | 0 | 0
Treated | 174 | 360 | 361 | 0 | 0
Completed | 0 | 202 | 202 | 0 | 0
Not Completed | 177 | 166 | 170 | 0 | 0
Not completed — Adverse Event | 14 | 27 | 60 | 0 | 0
Not completed — Pregnancy | 0 | 7 | 9 | 0 | 0
Not completed — Participant Defaulted | 11 | 40 | 36 | 0 | 0
Not completed — Lack of Efficacy | 11 | 64 | 30 | 0 | 0
Not completed — Death | 1 | 2 | 2 | 0 | 0
Not completed — Randomized, Not Treated | 3 | 8 | 11 | 0 | 0
Not completed — Protocol Violation | 2 | 18 | 22 | 0 | 0
Not completed — Terminated by sponsor | 135 | 0 | 0 | 0 | 0
Period: Between DB and OL Phase
Arm/Group | Maraviroc Once Daily + CBV (DB) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Maraviroc Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (SP)
Started | 0 | 202 | 202 | 0 | 0
Completed | 0 | 202 | 199 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0
Not completed — Did Not Enter Open-label Phase | 0 | 0 | 3 | 0 | 0
Period: Open-label (OL) Phase
Arm/Group | Maraviroc Once Daily + CBV (DB) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Maraviroc Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (SP)
Started | 0 | 202 | 199 | 130 | 0
Completed | 0 | 177 | 158 | 65 | 0
Not Completed | 0 | 25 | 41 | 65 | 0
Not completed — Adverse Event | 0 | 3 | 7 | 6 | 0
Not completed — Lack of Efficacy | 0 | 7 | 2 | 20 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 6 | 13 | 16 | 0
Not completed — Participant Defaulted | 0 | 6 | 16 | 20 | 0
Not completed — Death | 0 | 2 | 3 | 0 | 0
Period: Supplemental Phase (SP)
Arm/Group | Maraviroc Once Daily + CBV (DB) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Maraviroc Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (SP)
Started | 0 | 0 | 0 | 0 | 127
Completed | 0 | 0 | 0 | 0 | 94
Not Completed | 0 | 0 | 0 | 0 | 33
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 8
Not completed — Other | 0 | 0 | 0 | 0 | 22

BASELINE CHARACTERISTICS:
Groups:
- Efavirenz Once Daily + CBV (DB and OL): Placebo matched to maraviroc 300 mg tablet orally twice daily and efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, up to week 96 in DB phase. Efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily from Week 97 up to Week 240 in open-label (OL) phase.
- Total: Total of all reporting groups
Arm/Group | Maraviroc Once Daily + CBV (DB) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Total
Number analyzed (Participants) | 174 | 360 | 361 | 895
Age, Customized [Number; unit: participants]
  Less than 18 years | 0 | 0 | 0 | 0
  18 to 24 years | 17 | 24 | 25 | 66
  25 to 34 years | 47 | 147 | 120 | 314
  35 to 44 years | 73 | 117 | 141 | 331
  45 to 54 years | 29 | 56 | 55 | 140
  55 to 64 years | 7 | 14 | 15 | 36
  Greater than or equal to 65 years | 1 | 2 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 104 | 102 | 250
  Male | 130 | 256 | 259 | 645

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Viral Load of Less Than 400 Copies/Milliliter [Copies/mL] and Less Than 50 Copies/mL of Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) at Week 48 for Full Analysis Set (FAS) Population
Time Frame: Week 48
Population: FAS population included all the randomized participants who had taken at least 1 dose of the study medication. Missing data (MD) imputed as failure (F); that is, participants with missing data classified as not achieving the viral load criterion (MD=F).
Measure: Number; unit: Percentage of participants
Groups:
- Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL): Maraviroc 300 milligram (mg) tablet orally once daily in the evening along with placebo matched to maraviroc 300 mg tablet orally once daily in the morning and placebo matched to efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the DB phase prior to the termination of the treatment arm based on the recommendation of the DSMB following a planned interim analysis. Eligible participants then switched to open-label maraviroc 300 mg tablet orally twice daily co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily for the remainder of the study.
- Maraviroc Twice Daily + CBV (DB): Maraviroc 300 mg tablet orally twice daily and placebo matched to efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the DB phase.
- Efavirenz Once Daily + CBV (DB): Placebo matched to maraviroc 300 mg tablet orally twice daily and efavirenz 600 mg tablet orally once daily in the evening co-administered with combination therapy containing zidovudine 300 mg and lamivudine 150 mg (combivir [CBV]) tablet orally twice daily, during the DB phase.
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
Percentage of participants
  Less than 400 copies/mL | 61.5 | 70.6 | 73.1
  Less than 50 copies/mL | 55.8 | 65.3 | 69.3
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Treatment difference in percentages stratified by randomization strata (screening viral load and geographic region) was presented along with the lower bound of the 1-sided 97.5% confidence interval (CI) based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was greater than (>) -10%; Difference in Percentage = -3.0, 97.5% CI 1-sided [lower limit -9.5]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 50 copies/mL: Treatment difference in percentages stratified by randomization strata (screening viral load and geographic region) was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was > -10%; Difference in Percentage = -4.2, 97.5% CI 1-sided [lower limit -10.9]

2. Primary Outcome: Percentage of Participants With Viral Load of Less Than 400 Copies/mL and Less Than 50 Copies/mL of HIV-1 RNA at Week 48 for Per Protocol (PP) Population
Description: Percentage of participants with viral load of less than 400 copies/mL and less than 50 copies/mL of HIV-1 RNA were not analyzed for participants originally randomized to maraviroc once daily arm since after termination, focus was shifted from efficacy and safety to only safety as reflected in the abbreviated set of efficacy measures noted in the amended planned analysis.
Time Frame: Week 48
Population: Per protocol (PP) population included all randomized participants who had taken at least 1 dose of study medication, were treated for at least 14 days or discontinued before this time due to treatment failure, were >80% compliant with randomized treatment and had no violation of any inclusion or exclusion criteria, which affected efficacy. MD=F.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 360 | 361
Percentage of participants
  Less than 400 copies/mL | 75.00 | 78.27
  Less than 50 copies/mL | 70.00 | 74.44
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Treatment difference in percentage stratified by randomization strata (screening viral load and geographic region) was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was > -10%; Difference in Percentage = -4.1, 97.5% CI 1-sided [lower limit -10.5]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 50 copies/mL: Treatment difference in percentage stratified by randomization strata (screening viral load and geographic region) was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was > -10%; Difference in Percentage = -4.4, 97.5% CI 1-sided [lower limit -11.2]

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels of Less Than 400 Copies/mL and Less Than 50 Copies/mL at Week 48 Analyzed Using Logistic Regression
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
Percentage of participants
  Less than 400 copies/mL | 61.5 | 70.6 | 73.1
  Less than 50 copies/mL | 55.8 | 65.3 | 69.3
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Two-sided 95% CI was presented for the odds ratio between treatment groups. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (<100,000 or >=100,000), geographic region (Northern or Southern Hemisphere) as covariates was used. Odds ratio > 1 would favor maraviroc; Test type: Superiority or Other; p = 0.4485, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.64 to 1.22]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 50 copies/mL: Two-sided 95% CI was presented for the odds ratio between treatment groups. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (<100,000 or >=100,000), geographic region (Northern or Southern Hemisphere) as covariates were used. Odds ratio > 1 would favor maraviroc; Test type: Superiority or Other; p = 0.2724, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.61 to 1.15]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels of Less Than 400 Copies/mL and Less Than 50 Copies/mL at Week 96 Analyzed Using Logistic Regression
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
Percentage of participants
  Less than 400 copies/mL | 52.9 | 61.4 | 64.5
  Less than 50 copies/mL | 48.3 | 56.9 | 62.6
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Two-sided 95% CI was presented for the odds ratio between treatment groups. CIs were calculated using the Wald-approximation. Logistic model with treatment, screening HIV concentrations (<100,000 or >=100,000), geographic region (Northern or Southern Hemisphere) as covariates were used. Odds ratio > 1 would favor maraviroc; Test type: Superiority or Other; p = 0.3943, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.65 to 1.19]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.1289, Regression, Logistic; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.59 to 1.07]

5. Secondary Outcome: Change From Baseline in Log 10-transformed Plasma Viral Load (HIV-1 RNA) Levels at Week 48 and 96
Description: Change from baseline in log 10-transformed plasma viral load (HIV-1 RNA) levels (log10 copies/mL). Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and immediately pre-dose.
Time Frame: Baseline, Week 48, Week 96
Population: FAS population. Missing values for viral load at week 48 and 96 were imputed as baseline value for participants who discontinued and as last observation carried forward (LOCF) for participants who did not discontinue for maraviroc twice daily and efavirenz once daily arm and as LOCF for participants randomized to maraviroc once daily arm.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
log10 copies/mL
  Baseline | 4.899 (0.6273) | 4.851 (0.6511) | 4.857 (0.6156)
  Change at Week 48 | -2.665 (0.9454) | -2.240 (1.484) | -2.347 (1.455)
  Change at Week 96 | -2.565 (0.9731) | -1.961 (1.575) | -2.053 (1.564)
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at week 48: P-value was calculated using Analysis of Covariance (ANCOVA) with the model including treatment arm and, as covariates, the randomization strata (screening viral load and geographic region). The difference between the treatment least squares means (LS means) adjusted for the covariates was presented in addition to 2-sided 95% CI. Negative value would favor maraviroc; Test type: Superiority or Other; p = 0.2741, ANCOVA; LS Mean Difference = 0.118, 95% CI 2-sided [-0.094 to 0.329], Standard Error of Mean 0.1077
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at week 96: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Negative value would favor maraviroc; Test type: Superiority or Other; p = 0.3899, ANCOVA; LS Mean Difference = 0.100, 95% CI 2-sided [-0.128 to 0.328], Standard Error of Mean 0.1162

6. Secondary Outcome: Time-Averaged Difference (TAD) in log10-transformed HIV-1 RNA Levels
Description: TAD from baseline was calculated as area under the curve (AUC) of HIV-1 RNA load (log10 copies/mL) divided by time period minus baseline HIV-1 RNA load (log10 copies/mL). Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and immediately pre-dose. Data not analyzed for participants originally randomized to maraviroc once daily arm since after termination, focus was shifted from efficacy and safety to only safety as reflected in the abbreviated set of efficacy measures noted in the amended planned analysis.
Time Frame: Baseline up to Week 48 and Week 96
Population: FAS population included all the randomized participants who had taken at least 1 dose of the study medication. TAD imputed as 0 for participants who discontinued. TAD calculated using the last non-missing value prior to the analysis time point for participants with a missing value at the analysis time point but who had not discontinued.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 360 | 361
log10 copies/mL
  Week 48 | -2.152 (0.0713) | -2.262 (0.0714)
  Week 96 | -1.945 (0.0798) | -2.034 (0.0800)
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Week 48: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Negative value would favor maraviroc; Test type: Superiority or Other; p = 0.2693, ANCOVA; LS Mean Difference = 0.111, 95% CI 2-sided [-0.086 to 0.307], Standard Error of Mean 0.1002
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Week 96: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Negative value would favor maraviroc; Test type: Superiority or Other; p = 0.4270, ANCOVA; LS Mean Difference = 0.089, 95% CI 2-sided [-0.131 to 0.309], Standard Error of Mean 0.1121

7. Secondary Outcome: Change From Baseline in Lymphocyte Cluster of Differentiation 4 (CD4) Count at Week 48 and 96
Description: Baseline value calculated as the average of pre-dose measurements collected at screening and immediately pre-dose.
Time Frame: Baseline, Week 48, Week 96
Population: FAS population included all the randomized participants who had taken at least 1 dose of the study medication. 'N' (number of participants analyzed) signifies participants evaluable for this measure. Missing values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/µL)
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 360
cells per microliter (cells/µL)
  Baseline | 274.1 (175.45) | 264.70 (153.508) | 271.87 (133.491)
  Change at Week 48 | 172.50 (205.561) | 169.53 (134.409) | 143.52 (124.931)
  Change at Week 96 | 183.75 (166.454) | 206.31 (152.682) | 171.50 (149.163)
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at Week 48: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, baseline CD4 count and the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Positive value would favor maraviroc; Test type: Superiority or Other; p = 0.0075, ANCOVA; LS Mean Difference = 26.34, 95% CI 2-sided [7.04 to 45.63], Standard Error of Mean 9.827
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at Week 96: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, baseline CD4 count and the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Positive value would favor maraviroc; Test type: Superiority or Other; p = 0.0020, ANCOVA; LS Mean Difference = 35.44, 95% CI 2-sided [13.02 to 57.86], Standard Error of Mean 11.419

8. Secondary Outcome: Change From Baseline in Lymphocyte Cluster of Differentiation 8 (CD8) Count at Week 48 and 96
Description: Baseline value calculated as the average of pre-dose measurements collected at screening and immediately pre-dose. Change from baseline in lymphocyte CD8 count at Week 48 and 96 was not analyzed for participants originally randomized to maraviroc once daily arm since after termination, focus was shifted from efficacy and safety to only safety as reflected in the abbreviated set of efficacy measures noted in the amended planned analysis.
Time Frame: Baseline, Week 48, Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 360 | 360
cells/µL
  Baseline | 938.80 (503.392) | 935.78 (476.607)
  Change at Week 48 | 38.34 (397.503) | -126.83 (374.494)
  Change at Week 96 | 20.74 (412.081) | -150.27 (389.996)
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at Week 48: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, baseline CD8 count and the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Positive value would favor maraviroc; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = 166.29, 95% CI 2-sided [117.13 to 215.46], Standard Error of Mean 25.040
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Change at Week 96: P-value was calculated using ANCOVA with the model including treatment arm and, as covariates, baseline CD8 count and the randomization strata (screening viral load and geographic region). The difference between the treatment LS means adjusted for the covariates was presented in addition to 2-sided 95% CI. Positive value would favor maraviroc; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = 172.22, 95% CI 2-sided [122.21 to 222.23], Standard Error of Mean 25.471

9. Secondary Outcome: Time to Virologic Failure
Description: Time to virologic failure based on observed HIV-1 RNA levels and failure events (death;permanent discontinuation of drug;lost to follow-up [LTFU];new anti-retroviral drug added [except background drug change to drug of same class];or on open label for early non-response or rebound). Failure:at Time 0 if level not <400 copies/mL(2 consecutive visits) before events or last available visit;at time of earliest event if level <400 copies/mL(2 consecutive visits);failure if level >=400 copies/mL(2 consecutive visits) or 1 visit >=400 copies/mL followed by permanent discontinuation of drug or LTFU.
Time Frame: Week 48, Week 96
Population: FAS population; Data not analyzed for participants originally randomized to maraviroc once daily arm since after termination, focus was shifted from efficacy and safety to only safety as reflected in the abbreviated set of efficacy measures noted in the amended planned analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 360 | 361
days
  Week 48 | NA [354 to NA] — Median was not estimable because less than 50% of the participants experienced virological failure; upper confidence limit not estimable because the empirical distribution of the data rendered the algorithmic formula non-calculable. | NA [364 to NA] — Median was not estimable because less than 50% of the participants experienced virological failure; upper confidence limit not estimable because the empirical distribution of the data rendered the algorithmic formula non-calculable.
  Week 96 | NA [NA to NA] — Median was not estimable because less than 50% of the participants experienced virological failure; confidence limits not estimable because the empirical distribution of the data rendered the algorithmic formula non-calculable. | NA [691 to NA] — Median was not estimable because less than 50% of the participants experienced virological failure; upper confidence limit not estimable because the empirical distribution of the data rendered the algorithmic formula non-calculable.
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Week 48: P-value was calculated using Log rank test controlling for the effect of the randomization strata. Hazard ratio was calculated by fitting a Cox proportional hazards model including treatment group and the two randomization strata, HIV-1 RNA at screening and geographic region. Hazard ratio < 1 would favor maraviroc; Test type: Superiority or Other; p = 0.5874, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.83 to 1.45]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Week 96: P-value was calculated using Log rank test controlling for the effect of the randomization strata. Hazard ratio was calculated by fitting a Cox proportional hazards model including treatment group and the two randomization strata, HIV-1 RNA at screening and geographic region. Hazard ratio < 1 would favor maraviroc; Test type: Superiority or Other; p = 0.4811, Log Rank; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.86 to 1.40]

10. Secondary Outcome: Number of Participants Per Tropism Status at Baseline and at the Time of Treatment Failure Through Week 48
Description: Number of participants per tropism status (C-X-C chemokine receptor 5 {CCR5} [R5], C-X-C chemokine receptor type 4 {CXCR4} [X4], Dual/mixed [DM], or Non-reportable/Non-phenotypable [NR/NP]) at baseline and time of treatment failure analyzed through week 48 visit. Treatment failure: discontinuation due to insufficient clinical response. Tropism result was censored for participants with viral load <500 copies/mL at time of treatment failure categorized as below lower limit of quantification (BLQ). The assessment for time of treatment failure was defined as last on treatment assessment.
Time Frame: Baseline, time of failure through Week 48
Population: FAS population included all the randomized participants who had taken at least 1 dose of the study medication. 'N' (number of participants analyzed) is signifying those participants who experienced treatment failure, defined as discontinuation due to insufficient response and had tropism assessment at baseline.
Measure: Number; unit: participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 20 | 42 | 15
participants
  Baseline: R5; Treatment failure: R5 | 5 | 11 | 6
  Baseline: R5; Treatment failure: X4 | 0 | 0 | 0
  Baseline: R5; Treatment failure: DM | 3 | 10 | 0
  Baseline: R5; Treatment failure: NR/NP | 5 | 5 | 4
  Baseline: DM; Treatment failure: R5 | 0 | 1 | 0
  Baseline: DM; Treatment failure: X4 | 0 | 2 | 0
  Baseline: DM; Treatment failure: DM | 5 | 4 | 0
  Baseline: DM; Treatment failure: NR/NP | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Per Tropism Status at Baseline and at the Time of Treatment Failure Through Week 96
Description: Number of participants per tropism status (R5, X4, DM, or NR/NP) at baseline and time of treatment failure analyzed through week 96 visit. Treatment failure defined as insufficient clinical response. Tropism result was censored for participants with viral load <500 copies/mL at time of treatment failure categorized as BLQ. The assessment for time of treatment failure was defined as last on treatment assessment.
Time Frame: Baseline, time of failure through Week 96
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 27 | 54 | 23
participants
  Baseline: R5; Treatment failure: R5 | 9 | 14 | 10
  Baseline: R5; Treatment failure: X4 | 0 | 1 | 0
  Baseline: R5; Treatment failure: DM | 4 | 11 | 0
  Baseline: R5; Treatment failure: NR/NP | 6 | 7 | 5
  Baseline: DM; Treatment failure: R5 | 0 | 1 | 1
  Baseline: DM; Treatment failure: X4 | 0 | 2 | 0
  Baseline: DM; Treatment failure: DM | 5 | 4 | 0
  Baseline: DM; Treatment failure: NR/NP | 0 | 0 | 0
  Baseline: NR/NP; Treatment failure: R5 | 0 | 1 | 0
  Baseline: NR/NP; Treatment failure: X4 | 0 | 0 | 0
  Baseline: NR/NP; Treatment failure: DM | 0 | 0 | 0
  Baseline: NR/NP; Treatment failure: NR/NP | 0 | 1 | 0

12. Secondary Outcome: Number of Participants With Phenotypic Resistance at Time of Treatment Failure Through Week 48 and 96
Description: Phenotypic resistance to nucleoside reverse transcriptase inhibitors (NRTIs) and non-nucleoside reverse transcriptase inhibitors (NNRTIs) assessed at screening by Monogram Bioscience PhenoSense genotype (MBPSGT) assay, repeated if viral load >500 copies/mL at treatment failure through week 48, 96. Phenotypic resistance to maraviroc was assumed in maraviroc treatment failures with X4-using virus and in R5 maraviroc treatment failures using Monogram Bioscience PhenoSense Entry Assay. Phenotypic resistance to zidovudine, lamivudine, efavirenz and maraviroc at time of failure was summarized.
Time Frame: Screening, time of failure through Week 48, Week 96
Population: FAS population included all the randomized participants who had taken at least 1 dose of the study medication. 'n' is signifying those participants who experienced treatment failure, defined as discontinuation due to insufficient response at specified time points for each arm group respectively.
Measure: Number; unit: participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
participants
  Resistance to Zidovudine: Week 48 (n= 20, 43, 15) | 0 | 0 | 0
  Resistance to Lamivudine: Week 48 (n= 20, 43, 15) | 14 | 27 | 3
  Resistance to Efavirenz: Week 48 (n= 20, 43, 15) | 0 | 0 | 7
  Resistance to Maraviroc: Week 48 (n= 20, 43, 15) | NA — Data not summarized since treatment arm was stopped at Week 16 as it failed to meet pre-specified criteria. | 12 | NA — Data not summarized as maraviroc resistance was not relevant to efavirenz activity.
  Resistance to Zidovudine: Week 96 (n= 27, 55, 23) | 0 | 0 | 0
  Resistance to Lamivudine: Week 96 (n= 27, 55, 23) | 20 | 33 | 8
  Resistance to Efavirenz: Week 96 (n= 27, 55, 23) | 0 | 0 | 13
  Resistance to Maraviroc: Week 96 (n= 27, 55, 23) | NA — Data not summarized since treatment arm was stopped at Week 16 as it failed to meet pre-specified criteria. | NA — Data not summarized since Week 96 analysis included participants who experienced TLOVR defined virologic failure in addition to those with treatment failure. | NA — Data not summarized as maraviroc resistance was not relevant to efavirenz activity.

13. Secondary Outcome: Number of Participants With NRTI Associated Mutations at Time of Treatment Failure Through Week 48 and 96
Description: Genotypic resistance to NRTIs was assessed by identification of relevant mutations at screening using MBPSGT assay and repeated for all participants with HIV-1 viral load more than 500 copies/mL at treatment failure through week 48 and week 96. Following mutations associated with NRTIs were summarized at time of failure: Any zidovudine/lamivudine (Zid/Lam), Any thymidine analogue-associated mutation (TAM), methionine (M) to valine/isoleucine (V/I) substitution at residue (r) 184 (M184V/I), lysine (K) to arginine (R) substitution at residue 65 (K65R) and any other NRTI mutations.
Time Frame: Screening, time of failure through Week 48, Week 96
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
participants
  Any Zid/Lam Mutation: Week 48 (n= 20, 43, 15) | 14 | 27 | 3
  Any TAM Mutation: Week 48 (n= 20, 43, 15) | 1 | 6 | 0
  K65R Mutation: Week 48 (n= 20, 43, 15) | 0 | 1 | 0
  M184V/I Mutation: Week 48 (n= 20, 43, 15) | 14 | 27 | 3
  Other NRTI Mutation: Week 48 (n= 20, 43, 15) | 0 | 1 | 0
  Any Zid/Lam Mutation: Week 96 (n= 27, 55, 23) | 20 | 33 | 8
  Any TAM Mutation: Week 96 (n= 27, 55, 23) | 3 | 6 | 2
  K65R Mutation: Week 96 (n= 27, 55, 23) | 0 | 1 | 0
  M184V/I Mutation: Week 96 (n= 27, 55, 23) | 20 | 33 | 8
  Other NRTI Mutation: Week 96 (n= 27, 55, 23) | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With Efavirenz Associated Mutations at Time of Treatment Failure Through Week 48 and 96
Description: Genotypic resistance: mutations at screening by MBPSGT assay, repeated if viral load >500 copies/mL at treatment failure through week 48, 96. Efavirenz mutation:lysine to aspargine at r103(K103N);tyrosine to cysteine/isoleucine at r181(Y181C/I);tyrosine to cysteine/leucine/histidine at r188(Y188C/L/H);glycine to alanine/serine at r190(G190A/S);valine to alanine to r106(V106A);leucine to isoleucine at r100(L100I);alanine to glycine at r98(A98G);lysine to glutamic acid at r101(K101E);valine to isoleucine at r108(V108I);proline to histidine at r225(P225H);methionine to leucine at r230(M230L).
Time Frame: Screening, time of failure through Week 48, Week 96
Population: FAS population; n=participants with treatment failure at specified time points for each arm group respectively. Data not analyzed for participants originally randomized to maraviroc once daily arm since after termination focus shifted from efficacy, safety to only safety as reflected in abbreviated set of efficacy noted in amended planned analysis.
Measure: Number; unit: participants
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 360 | 361
participants
  L100I Mutation: Week 48 (n= 43, 15) | 0 | 0
  K103N Mutation: Week 48 (n= 43, 15) | 0 | 6
  V106M Mutation: Week 48 (n= 43, 15) | 0 | 0
  V108I Mutation: Week 48 (n= 43, 15) | 1 | 0
  Y181C/I Mutation: Week 48 (n= 43, 15) | 0 | 0
  Y188L Mutation: Week 48 (n= 43, 15) | 0 | 0
  G190S/A Mutation: Week 48 (n= 43, 15) | 0 | 1
  P225H Mutation: Week 48 (n= 43, 15) | 0 | 0
  L100I Mutation: Week 96 (n= 55, 23) | 0 | 0
  K103N Mutation: Week 96 (n= 55, 23) | 0 | 12
  V106M Mutation: Week 96 (n= 55, 23) | 0 | 1
  V108I Mutation: Week 96 (n= 55, 23) | 1 | 1
  Y181C/I Mutation: Week 96 (n= 55, 23) | 0 | 0
  Y188L Mutation: Week 96 (n= 55, 23) | 0 | 0
  G190S/A Mutation: Week 96 (n= 55, 23) | 0 | 2
  P225H Mutation: Week 96 (n= 55, 23) | 0 | 1

15. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels Less Than 50 Copies/mL at Week 48 and Week 96 by Overall Susceptibility Score (OSS) at Screening
Description: Association between baseline resistance and virological response was assessed as percentage of participants with HIV-1RNA levels less than 50 copies/mL by OSS at screening. OSS categorized as 0, 1, 2, >3 (maximum value of 6) and calculated as the sum of the net assessment of in-vitro phenotypic and genotypic susceptibility using a binary scoring system (0= resistant, 1= sensitive or susceptible) for each antiretroviral agent in OBT. Higher scores indicate greater susceptibility.
Time Frame: Baseline, Week 48, Week 96
Population: Data not analyzed because of insufficient diversity amongst participants with respect to baseline resistance due to the study entry criteria regarding baseline resistance.
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 0 | 0 | 0

16. Other Pre Specified Outcome: Percentage of Participants With Viral Load of Less Than 400 Copies/mL and Less Than 50 Copies/mL of HIV-1 RNA at Week 96
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 174 | 360 | 361
Percentage of participants
  Less than 400 copies/mL | 52.9 | 61.4 | 64.5
  Less than 50 copies/mL | 48.3 | 56.9 | 62.6
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Treatment difference in percentage stratified by randomization strata was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was greater than (>) -10%; Difference in Percentage = -3.2, 97.5% CI 1-sided [lower limit -10.2]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 50 copies/mL: Treatment difference in percentage stratified by randomization strata was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Step down procedure used to control for multiple comparisons; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower bound of the 1-sided 97.5% CI was > -10%; Difference in Percentage = -5.8, 97.5% CI 1-sided [lower limit -12.8]

17. Post Hoc Outcome: Percentage of Participants With HIV-1 RNA Levels of Less Than 400 Copies/mL and Less Than 50 Copies/mL at Week 48 for Enhanced Sensitivity Trofile Assay (ESTA) R5 Participants
Description: Percentage of participants with HIV-1 RNA levels of less than 400 copies/mL and less than 50 copies/mL were not analyzed for maraviroc once daily, then twice daily arm in order to avoid misinterpretation due to possible bias due to the fact that only a non-random sample of participants in the terminated arm were re-assayed with ESTA.
Time Frame: Week 48
Population: FAS population; 'N' number of participants analyzed included ESTA R5 participants who had R5 tropic virus by ESTA at screening. Missing data (MD) imputed as failure (F); that is, participants with missing data classified as not achieving the viral load criterion (MD=F).
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 311 | 303
Percentage of participants
  Less than 400 copies/mL | 73.3 | 72.3
  Less than 50 copies/mL | 68.5 | 68.3
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 400 copies/mL: Treatment difference in percentage stratified by randomization strata was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Due to its post-hoc nature, this analysis was considered descriptive only rather than inferential; Test type: Superiority or Other; Difference in Percentage = 0.6, 97.5% CI 1-sided [lower limit -6.4]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); Less than 50 copies/mL: Treatment difference in percentage stratified by randomization strata was presented along with the lower bound of the 1-sided 97.5% CI based on the normal approximation to the binomial distribution. Positive value would favor maraviroc. Due to its post-hoc nature, this analysis was considered descriptive only rather than inferential; Test type: Superiority or Other; Difference in Percentage = -0.2, 97.5% CI 1-sided [lower limit -7.4]

18. Post Hoc Outcome: Percentage of Participants With HIV-1 RNA Levels of Less Than 400 Copies/mL and Less Than 50 Copies/mL at Week 96 for Enhanced Sensitivity Trofile Assay (ESTA) R5 Participants
Description: as for outcome 17
Time Frame: Week 96
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc Twice Daily + CBV (DB) | Efavirenz Once Daily + CBV (DB)
Number analyzed (Participants) | 311 | 303
Percentage of participants
  Less than 400 copies/mL | 64.0 | 64.4
  Less than 50 copies/mL | 58.8 | 62.7
Statistical Analysis 1: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Difference in Percentage = -0.4, 97.5% CI 1-sided [lower limit -7.9]
Statistical Analysis 2: Comparison: Maraviroc Twice Daily + CBV (DB) vs Efavirenz Once Daily + CBV (DB); [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; Difference in Percentage = -3.9, 97.5% CI 1-sided [lower limit -11.5]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) | Maraviroc Twice Daily + CBV (DB and OL) | Efavirenz Once Daily + CBV (DB and OL) | Maraviroc Twice Daily + CBV (SP)
Serious Adverse Events (participants affected / at risk) | 47/174 | 77/360 | 82/361 | 4/127
Other Adverse Events (participants affected / at risk) | 151/174 | 319/360 | 327/361 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) (N=174) | Maraviroc Twice Daily + CBV (DB and OL) (N=360) | Efavirenz Once Daily + CBV (DB and OL) (N=361) | Maraviroc Twice Daily + CBV (SP) (N=127)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 6 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarciton (Cardiac disorders) | 0 | 2 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1 | 0 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Haematotympanum (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vertigo (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Diabetic eye disease (Eye disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 4 | 4 | 5 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 2 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Anal fistula infection (Infections and infestations) | 0 | 1 | 0 | 0
Anogenital warts (Infections and infestations) | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 3 | 3 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Cryptosporidiosis infection (Infections and infestations) | 1 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 2 | 2 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Neurosyphilis (Infections and infestations) | 0 | 1 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic inflamatory disease (Infections and infestations) | 0 | 0 | 1 | 0
Penile infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 5 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 2 | 3 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Sinobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 2 | 0
Syphilis (Infections and infestations) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Heart injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Human bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Multiple fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0
Gama-glutamytransferase increased (Investigations) | 1 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hoadgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 3 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 2 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 1 | 0
Dyspraxia (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalitis (Nervous system disorders) | 1 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Vascular demetia (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 5 | 8 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Drug dependence (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 2 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine cervical laceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug abuser (Social circumstances) | 1 | 0 | 0 | 0
Pregnancy of partner (Social circumstances) | 0 | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Finger amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc Once Daily + CBV (DB), Then Twice Daily + CBV (OL) (N=174) | Maraviroc Twice Daily + CBV (DB and OL) (N=360) | Efavirenz Once Daily + CBV (DB and OL) (N=361) | Maraviroc Twice Daily + CBV (SP) (N=127)
Anaemia (Blood and lymphatic system disorders) | 12 | 27 | 18 | 0
Conjunctivitis (Eye disorders) | 11 | 11 | 25 | 0
Abdominal distension (Gastrointestinal disorders) | 12 | 21 | 20 | 0
Abdominal pain (Gastrointestinal disorders) | 30 | 53 | 53 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 22 | 23 | 0
Constipation (Gastrointestinal disorders) | 13 | 37 | 20 | 0
Diarrhoea (Gastrointestinal disorders) | 46 | 90 | 111 | 0
Dyspepsia (Gastrointestinal disorders) | 9 | 26 | 38 | 0
Flatulence (Gastrointestinal disorders) | 10 | 26 | 13 | 0
Gastritis (Gastrointestinal disorders) | 5 | 16 | 22 | 0
Haemorrhoids (Gastrointestinal disorders) | 6 | 25 | 16 | 0
Nausea (Gastrointestinal disorders) | 60 | 138 | 132 | 0
Vomiting (Gastrointestinal disorders) | 28 | 53 | 61 | 0
Asthenia (General disorders) | 17 | 29 | 40 | 0
Chest pain (General disorders) | 6 | 17 | 25 | 0
Fatigue (General disorders) | 37 | 64 | 60 | 0
Influenza like illness (General disorders) | 14 | 21 | 22 | 0
Pyrexia (General disorders) | 16 | 21 | 30 | 0
Bronchitis (Infections and infestations) | 28 | 64 | 49 | 0
Gastroenteritis (Infections and infestations) | 10 | 27 | 33 | 0
Herpes zoster (Infections and infestations) | 4 | 18 | 16 | 0
Influenza (Infections and infestations) | 15 | 56 | 50 | 0
Nasopharyngitis (Infections and infestations) | 24 | 70 | 48 | 0
Pharyngitis (Infections and infestations) | 15 | 24 | 33 | 0
Sinusitis (Infections and infestations) | 4 | 29 | 28 | 0
Syphilis (Infections and infestations) | 10 | 16 | 13 | 0
Upper respiratory tract infection (Infections and infestations) | 32 | 82 | 78 | 0
Urinary tract infection (Infections and infestations) | 7 | 15 | 25 | 0
Alanine aminotransferase increased (Investigations) | 15 | 20 | 11 | 0
Aspartate aminotransferase increased (Investigations) | 12 | 13 | 12 | 0
Decreased appetite (Metabolism and nutrition disorders) | 18 | 34 | 36 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 37 | 30 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 44 | 44 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 16 | 22 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 29 | 28 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 27 | 23 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6 | 14 | 0
Dizziness (Nervous system disorders) | 25 | 62 | 116 | 0
Dysgeusia (Nervous system disorders) | 10 | 10 | 11 | 0
Headache (Nervous system disorders) | 44 | 109 | 105 | 0
Paraesthesia (Nervous system disorders) | 7 | 19 | 13 | 0
Somnolence (Nervous system disorders) | 6 | 18 | 13 | 0
Abnormal dreams (Psychiatric disorders) | 20 | 22 | 46 | 0
Anxiety (Psychiatric disorders) | 8 | 21 | 26 | 0
Depression (Psychiatric disorders) | 18 | 40 | 28 | 0
Insomnia (Psychiatric disorders) | 20 | 48 | 44 | 0
Sleep disorder (Psychiatric disorders) | 7 | 12 | 19 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 51 | 66 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 30 | 21 | 0
Eczema (Skin and subcutaneous tissue disorders) | 6 | 9 | 22 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 7 | 12 | 21 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 8 | 26 | 0
Rash (Skin and subcutaneous tissue disorders) | 25 | 38 | 56 | 0
Hypertension (Vascular disorders) | 6 | 25 | 23 | 0

LIMITATIONS AND CAVEATS:
Following DSMB decision to discontinue maraviroc 300 mg once daily, inferential statistical analyses was performed between maraviroc 300 mg twice daily and efavirenz 600 mg once daily only. Data at Week 24 was not analyzed as planned in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.